CLINICAL TRIAL: NCT02185898
Title: A Single-Center Evaluation of Environmental Emissions From Electronic Cigarettes and Tobacco-Burning Cigarettes
Brief Title: Evaluation of Environmental Emissions From Electronic Cigarettes and Tobacco-Burning Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R.J. Reynolds Vapor Company (Industry)
Collaborators: Covance (Industry); R.J. Reynolds Tobacco Company (Industry); MAS (Materials Analytical Services), LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CSD1302
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Smoking
Keywords: electronic cigarettes; e-cigarettes; combustible cigarettes; second-hand smoke; environmental tobacco smoke; tobacco-burning
MeSH Terms: conditions — Smoking; Vaping | interventions — Menthol; Nicotine; UBE2N protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Leading U.S. tobacco-burning non-menthol cigarette (Active Comparator): Leading U.S. non-menthol cigarette
  Interventions: Other: Leading U.S. non-menthol cigarette
- Leading U.S. tobacco-burning menthol cigarette (Active Comparator): Leading U.S. menthol cigarette
  Interventions: Other: Leading U.S. menthol cigarette
- Electronic cigarette #1 (Experimental): VUSE® (menthol flavor, 29 mg nicotine)
  Interventions: Other: Electronic cigarette #1
- Electronic cigarette #2 (Experimental): VUSE® (original flavor, 29 mg nicotine)
  Interventions: Other: Electronic cigarette #2
- Electronic cigarette #3 (Experimental): VUSE® (original flavor, 14 mg nicotine)
  Interventions: Other: Electronic cigarette #3
- U.S. Market-sample electronic cigarettes (two brands) (Experimental): blu™ (any variety) and NJOY® (any variety)
  Interventions: Other: U.S. Market-sample electronic cigarettes

INTERVENTIONS:
Other: Leading U.S. non-menthol cigarette — Tobacco-burning non-menthol cigarette
  Other Names: Marlboro Gold Pack Box
  Arms: Leading U.S. tobacco-burning non-menthol cigarette
Other: Leading U.S. menthol cigarette — Tobacco-burning menthol cigarette
  Other Names: Newport Box
  Arms: Leading U.S. tobacco-burning menthol cigarette
Other: Electronic cigarette #1 — Electronic cigarette
  Other Names: VUSE® Digital Vapor Cigarette (menthol flavor, 29 mg nicotine)
  Arms: Electronic cigarette #1
Other: Electronic cigarette #2 — Electronic cigarette
  Other Names: VUSE® Digital Vapor Cigarette (original flavor, 29 mg nicotine)
  Arms: Electronic cigarette #2
Other: Electronic cigarette #3 — Electronic cigarette
  Other Names: VUSE® Digital Vapor Cigarette (original flavor, 14 mg nicotine)
  Arms: Electronic cigarette #3
Other: U.S. Market-sample electronic cigarettes — Marketed electronic cigarettes
  Other Names: blu™ (any variety) and NJOY® (any variety)
  Arms: U.S. Market-sample electronic cigarettes (two brands)

SUMMARY:
This study will assess environmental emissions of selected compounds in a test chamber after cigarette smoking or e-cigarette vaping.

DETAILED DESCRIPTION:
Secondhand smoke is the aged and diluted combination of smoke exhaled by a smoker and sidestream smoke (smoke from the lit end of a cigarette). Electronic cigarettes are different from tobacco-burning cigarettes in that they produce vapor, not smoke. For consistency with common usage, secondhand smoke (SHS) refers to true secondhand smoke from cigarettes and secondhand vapor from e-cigarettes.

The goals of this study are to 1) increase understanding of the composition of SHS from e-cigarettes, 2) quantitatively compare the amount of SHS generated by e-cigarettes and a market sample of commercial e-cigarettes to leading brand styles of commercial tobacco-burning cigarettes, and 3) quantitate the emission factors of e-cigarettes including the market-sample e-cigarettes.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an Informed Consent Form (ICF) and complete questionnaires written in English.
2. Generally healthy males or females, 21 years of age or older at Screening.
3. Able to meet cohort-specific requirements as follows:

   Cohort 1 - Leading U.S. tobacco-burning non-menthol cigarette, and

   Cohort 2 - Leading U.S. tobacco-burning menthol cigarette:
   * self-reports at the Screening Visit smoking at least 5 cigarettes per day and inhaling the smoke, for at least 3 months prior to Screening
   * self-reports smoking Leading U.S. tobacco-burning non-menthol cigarette or Leading U.S. tobacco-burning menthol cigarette as usual brand (UB) cigarettes [UB cigarette is defined as the cigarette brand style currently smoked most frequently by the participant];

   Cohort 3 - Electronic cigarette #1 smokers, and

   Cohort 4 - Electronic cigarette #2 smokers:
   * self-reports at the Screening Visit smoking a non-menthol e-cigarette at least once per day, for at least 3 months prior to Screening;
   * willing to switch from using their current e-cigarette brand style to using a different e-cigarette brand style during the study;

   Cohort 5 - Electronic cigarette #3 smokers:
   * self-reports at the Screening Visit smoking a menthol e-cigarette at least once per day, for at least 3 months prior to Screening;
   * willing to switch from using their current e-cigarette brand style to using a different e-cigarette brand style during the study;

   Cohort 6 - U.S Market-sample electronic cigarette smokers:
   * self-reports at the Screening Visit smoking the selected U.S. market-sample e-cigarettes (menthol or non-menthol) at least once per day, for at least three months prior to Screening;
   * willing to continue exclusive use of their preferred style (flavor) of e-cigarette during the study.
4. Females of childbearing potential must be willing to use a form of contraception acceptable to the Investigator from the time of signing informed consent until study discharge or be surgically sterile for at least 90 days prior to enrollment;
5. Able to safely perform the required study procedures, as determined by the Investigator.

Exclusion Criteria:

1. Clinically significant or unstable/uncontrolled acute or chronic medical conditions at Screening, as determined by the Investigator, that would preclude a participant from participating safely in the study (e.g., hypertension, asthma, or other lung disease; cardiac disease; neurological disease; or psychiatric disorders) based on screening assessments such as safety labs and medical history or physical examination at Enrollment;
2. Self-reports or safety labs indicate diabetes;
3. At risk for heart disease, as determined by the Investigator;
4. Use of medicine for treatment of depression or asthma;
5. Systolic blood pressure of ≥150 mmHg or a diastolic blood pressure of ≥95 mmHg, measured after being seated for 5 minutes;
6. Postponing a decision to quit smoking (defined as planning a quit attempt within 30 days of the Screening Visit) to participate in this study;
7. Employed by a tobacco company, the study site, or environmental test chamber vendor;
8. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study;
9. History of claustrophobia;
10. Regularly exposed to solvent fumes or gasoline (e.g., painter, gas-station mini mart employee);
11. Determined by the Investigator to be inappropriate for this study, including a participant who is unable to communicate or unwilling to cooperate with the clinical staff.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To assess differences in levels of selected SHS constituents in an environmental test chamber after human smoking of e-cigarette #1, #2, and #3 compared to after human smoking of tobacco-burning cigarettes. | 2 weeks for participants in Cohorts 1 and 2; and approximately 4 weeks for participants in Cohorts 3, 4, and 5

SECONDARY OUTCOMES:
To determine selected SHS constituent emission factors for each tobacco-burning cigarette, each e-cigarette, and the market-sample e-cigarettes (collectively). | 2 weeks for participants in Cohorts 1, 2, and 6; and approximately 4 weeks for participants in Cohorts 3, 4, and 5
To assess the differences in levels of selected SHS constituents in an environmental test chamber after human smoking of e-cigarettes and tobacco-burning cigarettes compared to after a non-smoking blank condition. | 2 weeks for participants in Cohorts 1, 2, and 6; and approximately 4 weeks for participants in Cohorts 3, 4, and 5
To assess differences in levels of additional selected SHS constituents in an environmental test chamber after human smoking of e-cigarettes compared to after human smoking of tobacco-burning cigarettes. | 2 weeks for participants in Cohorts 1, 2, and 6; and approximately 4 weeks for participants in Cohorts 3, 4, and 5

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Segall, MD, CPI, Principal Investigator — Clinical Research Atlanta
Locations (1):
- Clinical Research Atlanta, Stockbridge, Georgia, United States

IPD SHARING:
Plan to Share IPD: No